CLINICAL TRIAL: NCT06275178
Title: Medical Thoracoscopy for Diagnosing Unexplained Pleural Effusion: a National Multicenter Retrospective Study
Status: Not yet recruiting | Type: Observational
Sponsor: China-Japan Friendship Hospital (Other)
Responsible Party: Principal Investigator, Gang Hou, Principal Investigator, China-Japan Friendship Hospital
Other Study IDs: ZRJY2021-BJ08-02-04
Record Dates: First submitted 2024-02-17; First posted 2024-02-23 (Actual); Last update posted 2024-02-23 (Actual); Status verified 2024-02

CONDITIONS: Pleural Effusion; Pleural Effusion, Malignant; Fibrinous Pleuritis
MeSH Terms: conditions — Pleural Effusion; Pleural Effusion, Malignant

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: Medical thoracoscopy — The included particpants are the patients with unexplained pleural effusion who underwent thoracoscopic or video-assisted thoracoscopic biopsy.

SUMMARY:
This study is a national multicenter retrospective study. Patients with unexplained pleural effusion who underwent thoracoscopic or video-assisted thoracoscopic biopsy for patients in recent 10 years were retrospectively collected from multiple centers to understand the proportion and final etiological composition of pleural effusion in China.

ELIGIBILITY:
Inclusion Criteria:

Patients with unexplained pleural effusion who underwent thoracoscopic or video-assisted thoracoscopic biopsy

Exclusion Criteria:

Patients who cannot obtain a final diagnosis

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with pleural effusion who underwent medical thoracoscopy were included in the study. Patients who could not obtain a final diagnosis were excluded from the study
Sampling Method: Non-Probability Sample
Enrollment: 5000 (Estimated)
Dates: Start 2024-03-20 (Estimated); Primary Completion 2024-12-24 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
The proportion of fibrinous pleurisy in Chinese population | December 31, 2024
  The proportion of fibrinous pleurisy in Chinese population